CLINICAL TRIAL: NCT04619394
Title: Analysis of the Effectiveness of Aquatic Exercise on the Static and Dynamic Balance in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: José M. Cancela (Other)
Responsible Party: Sponsor-Investigator, José M. Cancela, BENIGNA BLANCO NUÑEZ, University of Vigo
Organization: University of Vigo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: EACE01
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy; Aquatic Physical Exercise; Balance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (CG) (No Intervention): Control Group (CG): Formed by those pregnant women who do not perform any physical exercise, only the basic and instrumental activities of daily life (ABVD and AIVD respectively) and intensity of the physical labor load of very light to moderate. The period from 10-12 SG to 37-41 SG.
- Experimental Group 1 (GE1) (Active Comparator): Experimental Group 1 (GE1): Created for pregnant women who carry out their own program of each monitor in the different sports centers and public and private swimming pools in the South of the Autonomous Community of Galicia. These own programs will all have the same format: initial warm-up phase, main part of indicated and personalized exercises for pregnancies and final phase with a return to calm.
  Interventions: Other: Aquatic exercise - own monitors program
- Experimental Group 2 (GE2) (Active Comparator): Experimental Group 2 (GE2): In this third and last group, we incorporated the AIPAP program into the exclusive programs of each monitor in the various public and private sports centers and swimming pools in the South of the Autonomous Community of Galicia. The researcher trained in this method, together with the monitors who voluntarily wish to do so, will translate said format and program into their sessions.
  Interventions: Other: Aquatic exercise - AIPAP program

INTERVENTIONS:
Other: Aquatic exercise - own monitors program — Supervision of own exercises by the Monitor with its own program. Two weekly sessions, both aquatic in small glass and large. The activity carried out will be aerobic; They will work with their own body weight and the lightweight floating material they offer in these pools. Exercises will be carried out that favor flexibility, elasticity, resistance and the strengthening of the muscular ligaments. The intensity of the exercises will be moderate and adapted in each month of gestation. We will eliminate positions and exercises that overload the pregnant woman, avoiding possible injuries and obstetric alterations.
  The start of the program will be established in week 10-12 of the pregnancy and the end in week 37-41.
  The total number of sessions of the program will be from 25 to 31 (28 sessions of minimum compliance), with a frequency of 2 sessions per week. The duration of these will be 50 minutes and adherence to both experimental groups of ≥28 classes.
  Arms: Experimental Group 1 (GE1)
Other: Aquatic exercise - AIPAP program — Supervised by a midwife with AIPAP method. AIPAP method is divided into 10 sessions of 50 minutes that are repeated cyclically with a total of 120 exercises. The sessions are divided into 5 groups with different objectives: 2 sessions of aerobic capacity improvement, 2 sessions of strength improvement, 2 sessions of pelvic elasticity, 2 coordination sessions and the last 4 sessions of the previous ones.
  The beginning of the program will be established in week 10-12 of pregnancy and the end in week 37-41.
  The total number of sessions of the program will be 25-31 (28 sessions of minimum compliance), with a frequency of 2 sessions per week. The duration of these will be 50 minutes in both experimental groups. It will be necessary to obtain an adherence to both experimental groups of ≥28 classes.
  Arms: Experimental Group 2 (GE2)

SUMMARY:
Research about the balance in pregnant women who perform water exercise and those who do not engage in any type of sporting activity. The initial objectives are to know if there is an improvement in the balance in women who perform aquatic exercise reviewed at the end of pregnancy versus those who do not, through the use of a podiatric platform. This experimental randomized controlled study (RCT) will be carried out in sports centers and / or public or private municipal swimming pools in the south of Galicia The recruitment of passive pregnant women (control group) will be carried out in the health center of Pontevedra Virxe da Peregrina in the first visit to the midwife in the 10th and 12th week of gestation, while the recruitment of the active pregnant women (group experimental 1 and experimental group 2) in the teaching centers of the aquatic exercise sessions in the same weeks of gestation. The women of the three groups will have a low-risk normoevolutive pregnancy and will be studied in the first and third trimesters. The instruments that will be used to obtain data will be through an initial questionnaire, a platform and study of stability through the center of gravity and base of podiatric support. The plan for analyzing the data will be done through SPSS 17.0.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for inclusion of the sample are: 1. Women aged between 20 and 35 years since before 20 years and after 35 years it is associated with a greater maternal and perinatal risk.2. The intensity of the physical workload must be moderate to very light . 3. The gestational age (EG) in which they are captured must be delimited between 10 and 12 weeks of gestation (SG) without any obstetric risk or associated pathology, primiparous or multiparous.

Exclusion Criteria:

* Exclusion and withdrawal criteria. The exclusion criteria will be: 1. Present any type of absolute / relative obstetric contraindication. 2. Not to have notions of swimming. 3. Multiple pregnancies. 4. Pregnant women with cognitive / physical disability. 5. Present some diagnosed pathology that alters the normal balance as neurological, traumatological or podiatric diseases.

The appearance of any warning signs / symptoms such as vaginal bleeding, feeling light-headed or faint, difficulty breathing before doing exercise, chest pain, headache, muscle weakness, pain or swelling in the calves, Regular and painful contractions in the uterus and drip of fluid through the vagina, will imply the abandonment of the physical exercise program that was developing.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 75 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Balance | 24 weeks
  Balance analysis by force platform

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No